CLINICAL TRIAL: NCT00998764
Title: A Phase 3 Extension, Multicenter, Long Term Safety And Tolerability Trial Of Bapineuzumab (Aab 001, Eln115727) In Subjects With Alzheimer Disease Who Are Apolipoprotein E 4 Carriers And Participated In Study 3133k1-3001-us Or Study 3133k1-3001-ww.
Brief Title: A Long-Term Safety And Tolerability Extension Study Of Bapineuzumab In Alzheimer Disease Patients
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was terminated on August 6, 2012, because 2 large Phase 3 studies showed no clinical benefit. This decision was not based on any new safety concerns.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3133K1-3003; B2521004 (Other: Alias Study Number); 2009-015080-13 (EudraCT Number)
Record Dates: First submitted 2009-10-16; First posted 2009-10-20 (Estimated); Results first posted 2016-01-01 (Estimated); Last update posted 2016-01-01 (Estimated); Status verified 2015-11

CONDITIONS: Alzheimer Disease
Keywords: antibody; immunotherapy
MeSH Terms: conditions — Alzheimer Disease | interventions — bapineuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bapineuzumab 0.5 mg/kg (Experimental)
  Interventions: Drug: Bapineuzumab 0.5 mg/kg

INTERVENTIONS:
Drug: Bapineuzumab 0.5 mg/kg — I.V., 0.5 mg/kg, infusion every 13 weeks for a total of 16 infusions.
  Other Names: AAB-001

SUMMARY:
The purpose of this study is to assess the long-term safety and tolerability of bapineuzumab in subjects with Alzheimer Disease who participated in study 3133K1-3001(NCT00676143). Over 250 sites will participate in over 26 countries. Subjects will receive bapineuzumab. Each subject's participation will last approximately 4 years.

ELIGIBILITY:
Inclusion Criteria:

* Subject has completed study 3133K1-3001 (Week 78) and brain magnetic resonance imaging (MRI) scan consistent with the diagnosis of Alzheimer Disease
* Mini-Mental Status Examination (MMSE) >=10 at screening
* Caregiver able to attend all clinic visits with subject

Exclusion Criteria:

* Any medical or psychiatric contraindication or clinically significant abnormality that, in the investigator's judgment, will substantially increase the risk associated with the subject's participation in and completion of the study or could preclude the evaluation of the subject's response.
* Any significant brain MRI abnormality.
* Use of any investigational drugs or devices, other than bapineuzumab within the last 60 days prior to screening

Ages: 51 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 494 (Actual)
Dates: Start 2009-12; Primary Completion 2012-10 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (182):
- United States (65):
  - University Of Alabama at Birmingham, Birmingham, Alabama
  - UAB Center for Psychiatric Medicine, Birmingham, Alabama
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Alabama-Birmingham, Birmingham, Alabama
  - Dedicated Clinical Research, Goodyear, Arizona
  - Banner Alzheimer's Institute, Phoenix, Arizona
  - Banner Good Samaritan Medical Center (Imaging, Phoenix, Arizona
  - Jeffrey S. Gitt, Phoenix, Arizona
  - Hope Research Institute, Phoenix, Arizona
  - Clinical Trials, Inc., Little Rock, Arkansas
  - San Francisco Clinical Research Center, San Francisco, California
  - Alpine Clinical Research Center, Inc., Boulder, Colorado
  - Associated Neurologist, PC, Boulder, Colorado
  - Mile High Research Center, Denver, Colorado
  - Associated Neurologists of Southern Connecticut, P.C., Fairfield, Connecticut
  - Bendheim Infusion Center, Greenwich Hospital, Greenwich, Connecticut
  - Center for Healthy Aging, Greenwich Hospital, Greenwich, Connecticut
  - Research Center for Clinical Studies, Inc., Norwalk, Connecticut
  - JEM Research LLC, Atlantis, Florida
  - Medical Specialists of the Palm Beaches, Atlantis, Florida
  - Brain Matters Research, Delray Beach, Florida
  - Compass Research, LLC, Orlando, Florida
  - Palm Beach Neurological Center, Advanced Research Consultants, Inc., Palm Beach Gardens, Florida
  - Neurostudies, Inc, Port Charlotte, Florida
  - Southwest Florida Infusion Care, Inc., Port Charlotte, Florida
  - Roskamp Institute, Sarasota, Florida
  - USF Health Byrd Alzheimer's Institute, Tampa, Florida
  - Neuroscience Research Institute, LLC, Lawrenceville, Georgia
  - Neurostudies.net, Lawrenceville, Georgia
  - Alexian Brothers Neurosciences Institute Clinical Research, Elk Grove Village, Illinois
  - Southern Illinois University School of Medicine Department, Springfield, Illinois
  - Lake Charles Clinical Trials, Lake Charles, Louisiana
  - Neuroscience Research of the Berkshires, Pittsfield, Massachusetts
  - Springfield Neurology Associates, LLC, Springfield, Massachusetts
  - Michigan State University, East Lansing, Michigan
  - Neurological Research Center of Hattiesburg Clinic, Hattiesburg, Mississippi
  - The Center for Pharmaceutical Research, P.C., Kansas City, Missouri
  - Memory Enhancement Center of America, Inc., Eatontown, New Jersey
  - Alzheimer's Research Corp./Merician Institute for Aging, Paterson, New Jersey
  - Toms River X-Ray, CT & MRI, Toms River, New Jersey
  - MDR, Liverpool, New York
  - Neurological Care of Central New York, Liverpool, New York
  - Carolina Neuropsychological Services, Inc., Raleigh, North Carolina
  - Healthsouth Blue Ridge Surgery Center, Raleigh, North Carolina
  - Raleigh Neurology Associates, Raleigh, North Carolina
  - Wake Radiology Associates, Raleigh, North Carolina
  - Ohio State Unviersity, Columbus, Ohio
  - Summit Research Network(Oregon) Inc., Portland, Oregon
  - Providence Brain Institute-Cognitive Assessment Clinic, Portland, Oregon
  - Providence Brain Institute, Portland, Oregon
  - Abington Neurological Associates, Abington, Pennsylvania
  - Abington Neurological Assoc, Abington, Pennsylvania
  - Bington Memorial Hospital, Abington, Pennsylvania
  - Clinical Trial Center, LLC, Jenkintown, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Rhode Island Mood and Memory Research Institute, East Providence, Rhode Island
  - Medical University of South Carolina Hospitals and Clinics, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Medical University of South Carolina, North Charleston, South Carolina
  - Texas Neurology, P.A., Dallas, Texas
  - Innovative Clinical Trials, San Antonio, Texas
  - Integra Clinical Research, LLC, San Antonio, Texas
  - Vista Infusions, San Antonio, Texas
  - Inventive Infusion Solutions, San Antonio, Texas
- Hospital Italiano de Buenos Aires, Buenos Aires, Argentina
- Australia (8):
  - Gosford Hospital; Pharmacy Dept, Gosford, New South Wales
  - Hornsby Hospital, Hornsby, New South Wales
  - Royal Adelaide Memory Trials Centre, Adelaide, South Australia
  - Memory Unit 5C, Department of Neurology, Woodville South, South Australia
  - The Queen Elizabeth Hospital, Woodville South, South Australia
  - Heidelberg Repatriation Hospital, Heidelberg West, Victoria
  - Hollywood Hospital; Pharmacy Dept, Nedlands, Western Australia
  - The McCusker Foundation for Alzheimer's Disease Research, Nedlands, Western Australia
- Belgium (5):
  - ZNA Middelheim, Antwerp
  - AZ Sint-Jan Brugge-Oostende AV, Bruges
  - Cliniques Universitaires St Luc, Brussels
  - Universitair Ziekenhuis Gasthuisberg, Leuven
  - H.-Hartziekenhuis Roeselare-Menen, Roeselare
- Psicomedica Research Group, Santiago, Chile, Chile
- Finland (2):
  - Ita-Suomen Yliopisto, Kuopio
  - University of Turku/CRST, Turku
- France (18):
  - CHU de Dijon, Dijon, France
  - Hôpital Roger Salengro, Lille, France
  - Hôpital Pitié-Salpétrière, Paris, France
  - CHU Hôpital Pellegrin-Tripode, Bordeaux
  - Hopital Neurologique, Bron
  - CHU de Caen, Caen
  - Hôpitaux Civils de Colmar, Colmar
  - Hôpital la Timone, Marseille
  - CHU Hôpital Gui de Chaulliac, Montpellier
  - CHU Nord - Hôpital Guillaume et René Laënnec, Nantes - Saint Herblain
  - Hôpital Cimiez, Nice
  - CHU La Milétrie, Poitiers
  - C.H.U de Reims, Reims
  - Department de Radiologie et d'Imagerie Medicale, Hopital Pontchaillou, Rennes
  - CHRU Hôtel Dieu, Rennes
  - Centre Hospitalier Universitaire Charles Nicolle, Rouen
  - Hôpital Purpan, Toulouse
  - CHU Purpan - Hôpital Casselardit, Toulouse
- Italy (4):
  - Sezione di Neurologia - Dipartimento di Neuroscienze, Ancona
  - Dipartimento di Neuroscienze,, Catania
  - Fondazione IRCCS- Istituto Neurologico Carlo Besta, Milan
  - Unita' Operativa C - Riabilitazione Neurologica, Roma
- Japan (28):
  - Nagoya City University Hospital, Nagoya, Aichi-ken
  - Yachiyo Hospital, Aichi
  - Kashiwado Hospital, Chiba
  - National Hospital Organization Chiba-East Hospital, Chiba
  - Nippon Medical School Chiba Hokusoh Hospital, Chiba
  - National Hospital Organization Kokura Medical Center, Fukuoka
  - Maebashi Red Cross Hospital, Gunma
  - Gunma University Hospital, Gunma
  - Shinozuka Hospital, Gunma
  - National Hospital Organization Hiroshima-nishi Medical Ctr., Hiroshima
  - Kobe University Hospital, Hyōgo
  - Kagawa University Hospital, Kagawa
  - Nippon Medical School Musashi Kosugi Hospital, Kanagawa
  - Rakuwakai Otowa Hospital, Kyoto
  - National Hospital Organization Minami-Kyoto Hospital, Kyoto
  - National Hospital Organization Maizuru Medical Center, Kyoto
  - National Hospital Organization Matsumoto Medical Center, Nagano
  - National Hospital Organization Niigata National Hospital, Niigata
  - Okayama University Hospital, Okayama
  - National Hospital Organization Minami-Okayama Medical Center, Okayama
  - Osaka City University Hospital, Osaka
  - Kansai Medical University Takii Hospital, Osaka
  - Juntendo University Hospital, Tokyo
  - Juntendo Tokyo Koto Geriatric Medical Center, Tokyo
  - Tokyo Metropolitan Health and Med. Treatment Co. Ebara Hosp, Tokyo
  - Tokyo Medical University Hospital, Tokyo
  - Tokyo Medical University Hachioji Medical Center, Tokyo
  - National Hospital Organization Tokyo National Hospital, Tokyo
- Netherlands (4):
  - Geriatry, 's-Hertogenbosch
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - Vrije Universiteit Medisch Centrum, Amsterdam
  - Medisch Centrum Leeuwarden, Leeuwarden
- New Zealand (3):
  - The Memory Clinic Limited, Auckland
  - Christchurch Hospital, Christchurch
  - Signet Research, Christchurch
- Poland (6):
  - NZOZ Neuro-kard, Poznan, Poland
  - Pallmed Spolka z o.o., Bydgoszcz
  - MCD Voxel, Poznan
  - Pracownia Rezonansu Magnetycznego, Warsaw
  - SP ZOZ Szpital Wolski, Warsaw
  - Samodzielny Publiczny Centralny Szpital Kliniczny, Warsaw
- Portugal (3):
  - Hospitais Da Universidade De Coimbra, Coimbra, Coimbra District
  - Hospital Fernando da Fonseca, Amadora, Lisbon District
  - Hospital Santa Maria, Lisbon, Lisbon District
- Slovakia (2):
  - Univerzitna nemocnica Bratislava, Bratislava
  - Vseobecna nemocnica Rimavska Sobota, Rimavská Sobota
- South Africa (3):
  - Boithuso Caregivers, Johannesburg, Gauteng
  - The Osteoporosis and Memory Centre, Johannesburg, Gauteng
  - St Augustine's Medical Centre 2, Durban, KwaZulu-Natal
- Spain (14):
  - Hospital General Universitario de Elche, Elche, Alicante
  - Hospital Universitario Son Espases, Palma de Mallorca, Balearic Islands
  - CLONUS, Palma de Mallorca, Balearic Islands
  - Hospital del Mar, Barcelona, Barcelona
  - Fundacio ACE Institut Catala de Neurociences Aplicades, Barcelona, Barcelona
  - Clinica CIMA, Barcelona, Barcelona
  - Hospital Mutua de Terrasa, Terrassa, Barcelona
  - Hospital Divino Valles, Burgos, Burgos
  - Hospital Virgen del Puerto, Plasencia, Caceres
  - Hospital de la Princesa, Madrid, Madrid
  - Hospital Clinico San Carlos, Madrid, Madrid
  - Hospital Universitario La Paz, Madrid, Madrid
  - Hospital de la Princesa, Madrid
  - Hospital Universitario Virgen de la Arrixaca, Murcia
- Sweden (2):
  - Malmo University Hospital, Malmo
  - Minnes- och geriatrikmottagningen, Uppsala
- Memory Clinic Neuro-Psychologie Zentrum, Basel, Canton of Basel-City, Switzerland
- United Kingdom (12):
  - Memory Service North, Grenoside Grange Hospital, Grenoside, Sheffield
  - Llandough Hospital, Universtity Hospital of Wales, Cardiff, Wales
  - MAC UK Neuroscience Ltd., Bradford
  - Clinical Investigation and Research Unit (CIRU), Brighton
  - Glasgow Memory Clinic, Glasgow
  - Dept. of Neurosciences Charing Cross Hospital, London
  - The Doctors Laboratory Ltd., London
  - Newcastle General Hospital, Newcastle upon Tyne
  - Northampton General Hospital, Northampton
  - Royal Hallamshire Hospital, Sheffield
  - Victoria Hospital, Swindon
  - Alliance Medical, Wakefield

REFERENCES:
- [Derived] Ivanoiu A, Pariente J, Booth K, Lobello K, Luscan G, Hua L, Lucas P, Styren S, Yang L, Li D, Black RS, Brashear HR, McRae T. Long-term safety and tolerability of bapineuzumab in patients with Alzheimer's disease in two phase 3 extension studies. Alzheimers Res Ther. 2016 Jun 23;8(1):24. doi: 10.1186/s13195-016-0193-y. PMID 27334799
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3133K1-3003&StudyName=A%20Long-Term%20Safety%20And%20Tolerability%20Extension%20Study%20Of%20Bapineuzumab%20In%20Alzheimer%20Disease%20Patients

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 147 centers in 19 countries. The study was terminated early by the sponsor on 06 August 2012. Subjects who had not completed the final follow-up visit prior to 06 August 2012 were asked to complete an early termination visit.
Groups:
- Placebo/Bapineuzumab: Participants received placebo in the base study and bapineuzumab in this extension study. In this extension study bapineuzumab 0.5 mg/kg was administered by intravenous (IV) infusion approximately every 13 weeks up to week 195.
- Bapineuzumab/Bapineuzumab: Participants received bapinezumab in both the base and extension studies. In this extension study bapineuzumab 0.5 mg/kg was administered by IV infusion approximately every 13 weeks up to week 195.
Period: Overall Study
Arm/Group | Placebo/Bapineuzumab | Bapineuzumab/Bapineuzumab
Started | 216 | 276
Treated | 215 | 275
Completed | 0 | 2
Not Completed | 216 | 274
Not completed — Lack of Efficacy | 3 | 6
Not completed — Adverse Event | 17 | 12
Not completed — Withdrawal by Subject | 19 | 25
Not completed — Physician Decision | 3 | 3
Not completed — Death | 3 | 1
Not completed — Discontinuation of Study by Sponsor | 164 | 217
Not completed — Protocol Violation | 0 | 1
Not completed — Failed to Return | 1 | 1
Not completed — Lost to Follow-up | 1 | 1
Not completed — Loss of Caregiver | 0 | 3
Not completed — Other | 4 | 4
Not completed — Recurrent Episode of vasogenic edema | 1 | 0

BASELINE CHARACTERISTICS:
Population: The safety population included all participants who consented to participate in the extension and received at least one dose of the investigational product (in the extension study).
Groups:
- Placebo/Bapineuzumab: Participants received placebo in the base study and bapineuzumab in this extension study. In this extension study Bapineuzumab 0.5 mg/kg was administered by IV infusion approximately every 13 weeks up to week 195.
- Total: Total of all reporting groups
Arm/Group | Placebo/Bapineuzumab | Bapineuzumab/Bapineuzumab | Total
Number analyzed (Participants) | 215 | 275 | 490
Age, Continuous [Mean (Standard Deviation); unit: Years] | 71.4 (8.14) | 72.1 (7.47) | 71.8 (7.77)
Age, Customized [Number; unit: Participants]
  < 65 years | 44 | 42 | 86
  >= 65 years | 171 | 233 | 404
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 135 | 186 | 321
  Male | 80 | 89 | 169

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting a Serious Adverse Event
Description: Safety was measured according to standard adverse event collection as described in the Adverse Event Section of the Results. Complete tables of events are provided there.
Time Frame: Up to Week 195
Population: Safety population
Measure: Number; unit: Number of Participants
Groups:
- Bapineuzumab/Bapineuzumab: Participants received bapineuzumab in both the base and extension studies. In this extension study bapineuzumab 0.5 mg/kg was administered by IV infusion approximately every 13 weeks up to week 195.
Arm/Group | Placebo/Bapineuzumab | Bapineuzumab/Bapineuzumab
Number analyzed (Participants) | 215 | 275
Number of Participants | 35 | 33

2. Secondary Outcome: Change From Base Study Baseline in Alzheimer's Disease Assesment Scale-Cognitive Subscale (ADAS-Cog/11) at Weeks 13, 26, 39, 52 and 78
Description: The ADAS-Cog is a multi-item, objective measure of cognitive function. The scale evaluates memory, language, and praxis with items such as orientation, word recall, word recognition, object identification, comprehension, and the completion of simple tasks. Analysis of the ADAS-Cog for this study was based upon an 11 item score from the following items 1) word recall task, 2) naming objects and fingers, 3) following commands, 4)constructional praxis, 5) ideational praxis, 6) orientation, 7) word recognition, 8 remembering test instructions, 9) spoken language ability, 10) word finding difficulty in spontaneous speech, and 11) comprehension.This scale had to be administered by a trained and certified psychometric rater who did not have access to any information regarding adverse events experienced. The ADAS-Cog/11 ranged from 0 to 70 points, with higher scores indicating a greater degree of impairment. A negative change from baseline indicates a decrease in cognitive impairment.
Time Frame: Base Study Baseline, Weeks 13, 26, 39, 52 and 78
Population: The Modified Intent-to-Treat (mITT) Population was defined as all randomly assigned participants who received investigational product in the base study, had a baseline for the base study, had at least one valid post-baseline assessment of the ADAS-Cog and DAD total score in the base study and signed informed consent in the extension study.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo/Bapineuzumab | Bapineuzumab/Bapineuzumab
Number analyzed (Participants) | 199 | 256
Units on a scale
  Week 13 (N= 197, 253) | 5.53 (0.57) | 6.28 (0.50)
  Week 26 (N = 154, 221) | 7.41 (0.63) | 7.70 (0.54)
  Week 39 (N = 121, 184) | 8.83 (0.72) | 8.87 (0.61)
  Week 52 (N = 91, 139) | 10.12 (0.75) | 10.11 (0.63)
  Week 78 (N = 52, 80) | 13.91 (0.96) | 12.70 (0.80)
Statistical Analysis 1: Comparison: Placebo/Bapineuzumab vs Bapineuzumab/Bapineuzumab; Change from baseline in Alzheimer's Disease Assesment Scale-Cognitive Subscale (ADAS-Cog) at week 13; Test type: Superiority or Other; p = 0.324, Mixed Models Analysis; Mean Difference (Final Values) = 0.74, 95% CI 2-sided [-0.74 to 2.23]
Statistical Analysis 2: Comparison: Placebo/Bapineuzumab vs Bapineuzumab/Bapineuzumab; Change from baseline in Alzheimer's Disease Assesment Scale-Cognitive Subscale (ADAS-Cog) at week 26; Test type: Superiority or Other; p = 0.723, Mixed Models Analysis; Mean Difference (Final Values) = 0.29, 95% CI 2-sided [-1.33 to 1.92]
Statistical Analysis 3: Comparison: Placebo/Bapineuzumab vs Bapineuzumab/Bapineuzumab; Change from baseline in Alzheimer's Disease Assesment Scale-Cognitive Subscale (ADAS-Cog) at week 39; Test type: Superiority or Other; p = 0.966, Mixed Models Analysis; Mean Difference (Final Values) = 0.04, 95% CI 2-sided [-1.81 to 1.89]
Statistical Analysis 4: Comparison: Placebo/Bapineuzumab vs Bapineuzumab/Bapineuzumab; Change from baseline in Alzheimer's Disease Assesment Scale-Cognitive Subscale (ADAS-Cog) at week 52; Test type: Superiority or Other; p = 0.996, Mixed Models Analysis; Mean Difference (Final Values) = 0.00, 95% CI 2-sided [-1.93 to 1.92]
Statistical Analysis 5: Comparison: Placebo/Bapineuzumab vs Bapineuzumab/Bapineuzumab; Change from baseline in Alzheimer's Disease Assesment Scale-Cognitive Subscale (ADAS-Cog) at week 78; Test type: Superiority or Other; p = 0.336, Mixed Models Analysis; Mean Difference (Final Values) = -1.21, 95% CI 2-sided [-3.67 to 1.26]

3. Secondary Outcome: Change From Extension Study Baseline in ADAS-Cog/11 at Weeks 13, 26, 39, 52 and 78.
Description: The ADAS-Cog is a multi-item, objective measure of cognitive function. The scale evaluates memory, language, and praxis with items such as orientation, word recall, word recognition, object identification, comprehension, and the completion of simple tasks. Analysis of the ADAS-Cog for this study was based upon an 11 item score from the following items 1) word recall task, 2) naming objects and fingers, 3) following commands, 4)constructional praxis, 5) ideational praxis, 6) orientation, 7) word recognition, 8)remembering test instructions, 9) spoken language ability, 10) word finding difficulty in spontaneous speech, and 11) comprehension.This scale had to be administered by a trained and certified psychometric rater who did not have access to any information regarding adverse events experienced. The ADAS-Cog/11 ranged from 0 to 70 points, with higher scores indicating a greater degree of impairment. A negative change from baseline indicates a decrease in cognitive impairment.
Time Frame: Base Study Baseline, Weeks 13, 26, 39, 52 and 78
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo/Bapineuzumab | Bapineuzumab/Bapineuzumab
Number analyzed (Participants) | 199 | 256
Units on a scale
  Week 13 (N = 197, 253) | 0.89 (0.36) | 0.73 (0.32)
  Week 26 (N = 154, 221) | 2.87 (0.42) | 2.19 (0.35)
  Week 39 (N = 121, 184) | 4.26 (0.50) | 3.35 (0.42)
  Week 52 (N = 91, 139) | 5.42 (0.55) | 4.51 (0.45)
  Week 78 (N = 52, 80) | 9.21 (0.82) | 7.07 (0.66)
Statistical Analysis 1: Comparison: Placebo/Bapineuzumab vs Bapineuzumab/Bapineuzumab; Change from extension study baseline in ADAS-Cog at week 13; Test type: Superiority or Other; p = 0.737, Mixed Models Analysis; Mean Difference (Final Values) = -0.16, 95% CI 2-sided [-1.11 to 0.79]
Statistical Analysis 2: Comparison: Placebo/Bapineuzumab vs Bapineuzumab/Bapineuzumab; Change from extension study baseline in ADAS-Cog at week 26; Test type: Superiority or Other; p = 0.213, Mixed Models Analysis; Mean Difference (Final Values) = -0.68, 95% CI 2-sided [-1.76 to 0.40]
Statistical Analysis 3: Comparison: Placebo/Bapineuzumab vs Bapineuzumab/Bapineuzumab; Change from extension study baseline in ADAS-Cog at week 39; Test type: Superiority or Other; p = 0.168, Mixed Models Analysis; Mean Difference (Final Values) = -0.90, 95% CI 2-sided [-2.19 to 0.38]
Statistical Analysis 4: Comparison: Placebo/Bapineuzumab vs Bapineuzumab/Bapineuzumab; Change from extension study baseline in ADAS-Cog at week 52; Test type: Superiority or Other; p = 0.197, Mixed Models Analysis; Mean Difference (Final Values) = -0.91, 95% CI 2-sided [-2.30 to 0.48]
Statistical Analysis 5: Comparison: Placebo/Bapineuzumab vs Bapineuzumab/Bapineuzumab; Change from extension study baseline in ADAS-Cog at week 78; Test type: Superiority or Other; p = 0.044, Mixed Models Analysis; Mean Difference (Final Values) = -2.13, 95% CI 2-sided [-4.21 to 0.06]

4. Secondary Outcome: Change From Base Study Baseline in Disability Assessment for Dementia (DAD) Score at Weeks 13, 26, 39, 52 and 78.
Description: The DAD measures instrumental and basic activities of daily living in AD participants. The DAD is administered to the participant's caregiver in the form of an interview. The performance of basic activities of daily living is evaluated in 10 aspects including hygiene, dressing, continence, eating, meal preparation, telephoning, going on an outing, finance and correspondence, medications, leisure, and housework. The caregiver answers 40 questions as yes, no, or not applicable. A one-point score was assigned to each question if the answer is "yes" and a zero score was assigned if the answer is "no". For questions answered as "not applicable", no score will be assigned. The DAD total score was calculated as the total number of questions answered as "yes" divided by the total number of questions answered as "yes" or "no", times 100. The DAD score can range from 0 to 100, with higher scores indicating better function. A positive change indicates improvement from baseline.
Time Frame: Base Study Baseline, Weeks 13, 26, 39, 52 and 78
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Groups:
- Bapinezumab/Bapinezumab: Participants received bapinezumab in both the base and extension studies. In this extension study bapineuzumab 0.5 mg/kg was administered by IV infusion approximately every 13 weeks up to week 195.
Arm/Group | Placebo/Bapineuzumab | Bapinezumab/Bapinezumab
Number analyzed (Participants) | 199 | 256
Units on a scale
  Week 13 (N = 194, 247) | -12.33 (1.27) | 15.32 (1.11)
  Week 26 (N = 151, 222) | -15.37 (1.29) | -18.04 (1.11)
  Week 39 (N = 119, 180) | -17.74 (1.47) | -21.33 (1.24)
  Week 52 (N = 89, 137) | -20.96 (1.65) | -22.72 (1.36)
  Week 78 (N = 50, 81) | -26.33 (2.18) | -29.11 (1.75)
Statistical Analysis 1: Comparison: Placebo/Bapineuzumab vs Bapinezumab/Bapinezumab; Change from base study baseline in DAD score at Week 13; Test type: Superiority or Other; p = 0.077, Mixed Models Analysis; Mean Difference (Final Values) = -2.99, 95% CI 2-sided [-6.30 to 0.33]
Statistical Analysis 2: Comparison: Placebo/Bapineuzumab vs Bapinezumab/Bapinezumab; Change from base study baseline in DAD score at Week 26; Test type: Superiority or Other; p = 0.117, Mixed Models Analysis; Mean Difference (Final Values) = -2.67, 95% CI 2-sided [-6.02 to 0.67]
Statistical Analysis 3: Comparison: Placebo/Bapineuzumab vs Bapinezumab/Bapinezumab; Change from base study baseline in DAD score at Week 39; Test type: Superiority or Other; p = 0.063, Mixed Models Analysis; Mean Difference (Final Values) = -3.60, 95% CI 2-sided [-7.38 to 0.19]
Statistical Analysis 4: Comparison: Placebo/Bapineuzumab vs Bapinezumab/Bapinezumab; Change from base study baseline in DAD score at Week 52; Test type: Superiority or Other; p = 0.412, Mixed Models Analysis; Mean Difference (Final Values) = -1.75, 95% CI 2-sided [-5.95 to 2.44]
Statistical Analysis 5: Comparison: Placebo/Bapineuzumab vs Bapinezumab/Bapinezumab; Change from base study baseline in DAD score at Week 78; Test type: Superiority or Other; p = 0.321, Mixed Models Analysis; Mean Difference (Final Values) = -2.78, 95% CI 2-sided [-8.28 to 2.73]

5. Secondary Outcome: Change From Extension Study Baseline in Disability Assessment for Dementia (DAD) Score at Weeks 13, 26, 39, 52 and 78.
Description: as for outcome 4
Time Frame: Base Study Baseline, Weeks 13, 26, 39, 52 and 78
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on scale
Arm/Group | Placebo/Bapineuzumab | Bapinezumab/Bapinezumab
Number analyzed (Participants) | 199 | 256
Units on scale
  Week 13 (N = 194, 247) | -2.63 (0.83) | -3.71 (0.73)
  Week 26 (N = 151, 222) | -5.76 (1.01) | -6.46 (0.86)
  Week 39 (N = 119, 180) | -8.17 (1.22) | -9.72 (1.02)
  Week 52 (N = 89, 137) | -11.82 (1.34) | -11.11 (1.10)
  Week 78 (N = 50, 81) | -17.34 (1.94) | -17.48 (1.56)
Statistical Analysis 1: Comparison: Placebo/Bapineuzumab vs Bapinezumab/Bapinezumab; Change from extension study baseline in DAD score at Week 13; Test type: Superiority or Other; p = 0.329, Mixed Models Analysis; Mean Difference (Final Values) = -1.08, 95% CI 2-sided [-3.24 to 1.09]
Statistical Analysis 2: Comparison: Placebo/Bapineuzumab vs Bapinezumab/Bapinezumab; Change from extension study baseline in DAD score at Week 26; Test type: Superiority or Other; p = 0.601, Mixed Models Analysis; Mean Difference (Final Values) = -0.70, 95% CI 2-sided [-3.31 to 1.92]
Statistical Analysis 3: Comparison: Placebo/Bapineuzumab vs Bapinezumab/Bapinezumab; Change from extension study baseline in DAD score at Week 39; Test type: Superiority or Other; p = 0.328, Mixed Models Analysis; Mean Difference (Final Values) = -1.55, 95% CI 2-sided [-4.67 to 1.56]
Statistical Analysis 4: Comparison: Placebo/Bapineuzumab vs Bapinezumab/Bapinezumab; Change from extension study baseline in DAD score at Week 52; Test type: Superiority or Other; p = 0.680, Mixed Models Analysis; Mean Difference (Final Values) = 0.71, 95% CI 2-sided [-2.70 to 4.13]
Statistical Analysis 5: Comparison: Placebo/Bapineuzumab vs Bapinezumab/Bapinezumab; Change from extension study baseline in DAD score at Week 78; Test type: Superiority or Other; p = 0.954, Mixed Models Analysis; Mean Difference (Final Values) = -0.14, 95% CI 2-sided [-5.05 to 4.77]

6. Secondary Outcome: Change From Base Study Baseline in Neuropsychiatric Inventory (NPI) Score at Weeks 26, 52 and 78.
Description: NPI:12-domain caregiver assessment of behavioral disturbances occurring in dementia: delusions, hallucinations, agitation/ aggression, depression/dysphoria, anxiety, elation/euphoria, apathy/ indifference, disinhibition, irritability/lability, motor disturbance, appetite/eating, nighttime behavior. Severity(1=Mild to 3=Severe),frequency (1=occasionally to 4=very frequently) scales recorded for each domain; frequency*severity=each domain score(range 0-12). The NPI total score ranges from 0 to 144 with higher NPI scores indicate greater impairment. A negative change indicates improvement from baseline.
Time Frame: Base Study Baseline, Weeks 26, 52 and 78
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo/Bapineuzumab | Bapinezumab/Bapinezumab
Number analyzed (Participants) | 199 | 256
Units on a scale
  Week 26 (N = 176, 240) | 2.84 (0.97) | 2.95 (0.83)
  Week 52 (N = 110, 163) | 4.32 (0.96) | 3.52 (0.80)
  Week 78 (N = 51, 81) | 6.95 (1.70) | 4.93 (1.36)
Statistical Analysis 1: Comparison: Placebo/Bapineuzumab vs Bapinezumab/Bapinezumab; Change from base study baseline in NPI score at week 26; Test type: Superiority or Other; p = 0.931, Mixed Models Analysis; Mean Difference (Final Values) = 0.11, 95% CI 2-sided [-2.40 to 2.62]
Statistical Analysis 2: Comparison: Placebo/Bapineuzumab vs Bapinezumab/Bapinezumab; Change from base study baseline in NPI score at week 52; Test type: Superiority or Other; p = 0.524, Mixed Models Analysis; Mean Difference (Final Values) = -0.80, 95% CI 2-sided [-3.26 to 1.67]
Statistical Analysis 3: Comparison: Placebo/Bapineuzumab vs Bapinezumab/Bapinezumab; Change from base study baseline in NPI score at week 78; Test type: Superiority or Other; p = 0.353, Mixed Models Analysis; Mean Difference (Final Values) = -2.03, 95% CI 2-sided [-6.32 to 2.27]

7. Secondary Outcome: Change From Extension Study Baseline in NPI Score at Weeks 26, 52 and 78.
Description: as for outcome 6
Time Frame: Base Study Baseline, Weeks 26, 52 and 78
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo/Bapineuzumab | Bapinezumab/Bapinezumab
Number analyzed (Participants) | 199 | 256
Units on a scale
  Week 26 (N = 176, 240) | 2.17 (0.86) | 1.47 (0.73)
  Week 52 (N = 110, 163) | 3.82 (0.95) | 1.98 (0.79)
  Week 78 (N = 51, 81) | 6.60 (1.69) | 3.29 (1.35)
Statistical Analysis 1: Comparison: Placebo/Bapineuzumab vs Bapinezumab/Bapinezumab; Change from extension study baseline in NPI score at week 26; Test type: Superiority or Other; p = 0.531, Mixed Models Analysis; Mean Difference (Final Values) = -0.71, 95% CI 2-sided [-2.92 to 1.51]
Statistical Analysis 2: Comparison: Placebo/Bapineuzumab vs Bapinezumab/Bapinezumab; Change from extension study baseline in NPI score at week 52; Test type: Superiority or Other; p = 0.137, Mixed Models Analysis; Mean Difference (Final Values) = -1.84, 95% CI 2-sided [-4.28 to 0.59]
Statistical Analysis 3: Comparison: Placebo/Bapineuzumab vs Bapinezumab/Bapinezumab; Change from extension study baseline in NPI score at week 78; Test type: Superiority or Other; p = 0.128, Mixed Models Analysis; Mean Difference (Final Values) = -3.32, 95% CI 2-sided [-7.60 to 0.96]

8. Secondary Outcome: Change From Base Study Baseline in Mini-mental State Examination (MMSE) Score at Weeks 6, 19, 32, 45 and 78.
Description: MMSE measured general cognitive functioning: orientation, memory, attention, concentration, naming, repetition, comprehension, and ability to create a sentence and to copy two intersecting polygons. The MMSE total score can range from 0 to 30, with lower scores indicating a greater degree of impairment. A positive change indicates improvement from baseline.
Time Frame: Base Study Baseline, Weeks 6, 19, 32, 45 and 78
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo/Bapineuzumab | Bapinezumab/Bapinezumab
Number analyzed (Participants) | 199 | 256
Units on a scale
  Week 6 (N= 197, 255) | -2.61 (0.22) | -2.55 (0.19)
  Week 19 (N = 184, 241) | -3.13 (0.22) | -3.01 (0.19)
  Week 32 (N = 141, 204) | -3.75 (0.24) | -3.65 (0.20)
  Week 45 (N = 117, 171) | -4.44 (0.26) | -4.26 (0.21)
  Week 78 (N = 65, 94) | -5.50 (0.32) | -5.54 (0.26)
Statistical Analysis 1: Comparison: Placebo/Bapineuzumab vs Bapinezumab/Bapinezumab; Change from base study baseline in MMSE score at Week 6; Test type: Superiority or Other; p = 0.811, Mixed Models Analysis; Mean Difference (Final Values) = 0.07, 95% CI 2-sided [-0.49 to 0.63]
Statistical Analysis 2: Comparison: Placebo/Bapineuzumab vs Bapinezumab/Bapinezumab; Change from base study baseline in MMSE score at Week 19; Test type: Superiority or Other; p = 0.681, Mixed Models Analysis; Mean Difference (Final Values) = 0.12, 95% CI 2-sided [-0.45 to 0.69]
Statistical Analysis 3: Comparison: Placebo/Bapineuzumab vs Bapinezumab/Bapinezumab; Change from extension study baseline in MMSE score at Week 32; Test type: Superiority or Other; p = 0.742, Mixed Models Analysis; Mean Difference (Final Values) = 0.10, 95% CI 2-sided [-0.51 to 0.72]
Statistical Analysis 4: Comparison: Placebo/Bapineuzumab vs Bapinezumab/Bapinezumab; Change from extension study baseline in MMSE score at Week 45; Test type: Superiority or Other; p = 0.598, Mixed Models Analysis; Mean Difference (Final Values) = 0.18, 95% CI 2-sided [-0.48 to 0.83]
Statistical Analysis 5: Comparison: Placebo/Bapineuzumab vs Bapinezumab/Bapinezumab; Change from extension study baseline in MMSE score at Week 78; Test type: Superiority or Other; p = 0.922, Mixed Models Analysis; Mean Difference (Final Values) = -0.04, 95% CI 2-sided [-0.85 to 0.77]

9. Secondary Outcome: Change From Extension Study Baseline in MMSE Score at Weeks 6, 19, 32, 45 and 78.
Description: as for outcome 8
Time Frame: Base Study Baseline, Weeks 6, 19, 32, 45 and 78
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo/Bapineuzumab | Bapinezumab/Bapinezumab
Number analyzed (Participants) | 199 | 256
Units on a scale
  Week 6 (N = 195, 255) | -0.67 (0.19) | -0.26 (0.16)
  Week 19 (N = 182, 241) | -1.16 (0.21) | -0.69 (0.18)
  Week 32 (N = 140, 204) | -1.85 (0.24) | -1.40 (0.20)
  Week 45 (N = 116, 171) | -2.57 (0.28) | -2.05 (0.24)
  Week 78 (N = 64, 94) | -3.69 (0.39) | -3.42 (0.32)
Statistical Analysis 1: Comparison: Placebo/Bapineuzumab vs Bapinezumab/Bapinezumab; Change from extension study baseline in MMSE score at Week 6; Test type: Superiority or Other; p = 0.099, Mixed Models Analysis; Mean Difference (Final Values) = 0.41, 95% CI 2-sided [-0.08 to 0.90]
Statistical Analysis 2: Comparison: Placebo/Bapineuzumab vs Bapinezumab/Bapinezumab; Change from extension study baseline in MMSE score at Week 19; Test type: Superiority or Other; p = 0.089, Mixed Models Analysis; Mean Difference (Final Values) = 0.47, 95% CI 2-sided [-0.07 to 1.01]
Statistical Analysis 3: Comparison: Placebo/Bapineuzumab vs Bapinezumab/Bapinezumab; Change from extension study baseline in MMSE score at Week 32; Test type: Superiority or Other; p = 0.152, Mixed Models Analysis; Mean Difference (Final Values) = 0.45, 95% CI 2-sided [-0.17 to 1.08]
Statistical Analysis 4: Comparison: Placebo/Bapineuzumab vs Bapinezumab/Bapinezumab; Change from extension study baseline in MMSE score at Week 45; Test type: Superiority or Other; p = 0.160, Mixed Models Analysis; Mean Difference (Final Values) = 0.52, 95% CI 2-sided [-0.21 to 1.25]
Statistical Analysis 5: Comparison: Placebo/Bapineuzumab vs Bapinezumab/Bapinezumab; Change from extension study baseline in MMSE score at Week 78; Test type: Superiority or Other; p = 0.603, Mixed Models Analysis; Mean Difference (Final Values) = 0.26, 95% CI 2-sided [-0.73 to 1.26]

ADVERSE EVENTS:
Time Frame: 3 years
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Placebo/Bapineuzumab | Bapineuzumab/Bapineuzumab
Serious Adverse Events (participants affected / at risk) | 35/215 | 33/275
Other Adverse Events (participants affected / at risk) | 57/215 | 45/275
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo/Bapineuzumab (N=215) | Bapineuzumab/Bapineuzumab (N=275)
Aortic valve stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular block (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Mitral valve disease (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 4 (4)
Asthenia (General disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1)
Gait disturbance (General disorders) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (2) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Gastritis viral (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Peritonsillar abscess (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (1)
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Forearm fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 1 (1)
Cerebellar infarction (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral microhaemorrhage (Nervous system disorders) | 2 (2) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 1 (1) | 2 (2)
Epilepsy (Nervous system disorders) | 3 (3) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 1 (1)
Lacunar infarction (Nervous system disorders) | 1 (1) | 0 (0)
Lumbar radiculopathy (Nervous system disorders) | 0 (0) | 1 (1)
Multiple system atrophy (Nervous system disorders) | 0 (0) | 1 (1)
Partial seizures (Nervous system disorders) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 2 (2) | 0 (0)
Vasogenic cerebral oedema (Nervous system disorders) | 6 (6) | 2 (2)
Aggression (Psychiatric disorders) | 1 (1) | 2 (2)
Agitation (Psychiatric disorders) | 1 (1) | 2 (2)
Confusional state (Psychiatric disorders) | 0 (0) | 2 (2)
Delusion (Psychiatric disorders) | 0 (0) | 1 (1)
Hallucination (Psychiatric disorders) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1)
Mood swings (Psychiatric disorders) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1)
Incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Peripheral artery stenosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo/Bapineuzumab (N=215) | Bapineuzumab/Bapineuzumab (N=275)
Diarrhoea (Gastrointestinal disorders) | 12 (12) | 10 (13)
Cerebral microhaemorrhage (Nervous system disorders) | 18 (22) | 15 (16)
Headache (Nervous system disorders) | 16 (29) | 8 (8)
Vasogenic cerebral oedema (Nervous system disorders) | 17 (24) | 8 (8)
Anxiety (Psychiatric disorders) | 11 (13) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.